CLINICAL TRIAL: NCT06995014
Title: Retrieval-based Word Learning in Developmental Language Disorder: Adaptive Retrieval Schedule
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Laurence Leonard, Professor, Purdue University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1603017480D; R01DC014708 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Developmental Language Disorder; Specific Language Impairment; Language Development
Keywords: Word learning; Word retrieval; Preschool-aged children
MeSH Terms: conditions — Language Development Disorders; Specific Language Disorder

STUDY DESIGN:
Intervention Model Description: Within-participant design in which each child learns words under two conditions. The clinical group (children with DLD) is compared to the control group (children with Typical development) on these two word learning conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Developmental Language Disorder (Experimental): These children have a significant delay in language development in the absence of hearing impairment, cognitive delay, autism, or neurological injury/disease.
  Interventions: Behavioral: Retrieval-based word learning: Standard retrieval practice schedule; Behavioral: Retrieval-based word learning: Adaptive retrieval practice schedule
- Children With Typical Language Development (Experimental): Children whose language development is as expected for their age.
  Interventions: Behavioral: Retrieval-based word learning: Standard retrieval practice schedule; Behavioral: Retrieval-based word learning: Adaptive retrieval practice schedule

INTERVENTIONS:
Behavioral: Retrieval-based word learning: Standard retrieval practice schedule — Novel nouns and their meanings are practiced on 2 consecutive days. At the beginning of each learning session, a retrieval trial will immediately follow hearing the word and what it likes (a study trial). In the standard condition, the remaining retrieval trials for each word will be spaced - occurring only after 3 other words have intervened. This practice schedule is repeated the next day (Day 2).
Behavioral: Retrieval-based word learning: Adaptive retrieval practice schedule — Novel nouns and their meanings are practiced on 2 consecutive days. At the beginning of each learning session, a retrieval trial will immediately follow hearing the word and what it likes (a study trial). For the remainder of the session, there will be spaced retrieval trials for each word - occurring after 3 words have intervened. In the Adaptive condition, children will have additional retrieval opportunities throughout. These will be provided whenever the child does not remember the word form, whether it is an immediate (initial) or space retrieval trial. This practice schedule is repeated the next day (Day 2).

SUMMARY:
Children with developmental language disorder (DLD; also referred to as specific language impairment) experience a significant deficit in language ability that is longstanding and harmful to the children's academic, social, and eventual economic wellbeing. Word learning is one of the principal weaknesses in these children. This project focuses on the word learning abilities of four- and five-year-old children with DLD. The goal of the project is to determine whether special benefits accrue when these children must frequently recall newly introduced words during the course of learning. In the current study, the investigators compare a "standard" repeated spaced retrieval schedule, with fixed spacing between hearing a word and attempting to retrieve it, to an "adaptive" repeated spaced retrieval schedule in which opportunities to retrieve a given word are tailored to the individual child's current knowledge state. The goal of the study is to determine whether the adaptive schedule can increase children's absolute levels of learning while maintaining the advantages of repeated spaced retrieval.

DETAILED DESCRIPTION:
Developmental Language Disorder (DLD) affects language learning in an estimated 7% of children. Although much of the research literature has emphasized difficulties learning grammar, children with DLD also have major deficits in vocabulary. In recent work, the investigators have been examining the benefit of retrieval practice to enhance word learning and retention in preschoolers with DLD. The rationale behind this work is grounded in the growing literature in the field of cognitive psychology which shows that repeated practice in retrieving information results in greater long-term retention than continuous study of that information without opportunities for retrieval. In addition, retrieval practice that occurs after a delay-or "spacing" between study of a word and subsequent recall attempts-can lead to stronger effects.

Despite the growing evidence that repeated spaced retrieval (RSR) results in greater word learning for preschoolers with DLD, much remains to be learned. One important question concerns the absolute level of learning achieved through RSR. These investigators have found that, in the more optimal condition of RSR, these children's ability to recall new word forms (i.e., recall the phonetic form of the word such as /pobɪk/) is still low, despite being higher than recall in the comparison conditions. The main obstacle appeared to be initial word form encoding during the learning period. Longer-term retention was less of a problem, i.e., those words children could recall immediately after the learning period were also recalled one week later. In the current study, the investigators seek to improve word form recall through modifications that may improve this initial encoding. The principal means by which this study will attempt to improve encoding and, as a result, subsequent recall, is through an adaptive retrieval schedule, described below.

Sixteen children with DLD will be recruited for this study along with 16 children with typical language development (TD) matched on chronological age. Using a within-subjects design, children will learn eight novel verbs, four at a time. Each set of four will be learned over two consecutive days, with one block of four in the standard RSR condition and the other block in the adaptive RSR condition. The referents for these novel words will be photos of unfamiliar plants and animals, presented on a laptop screen. Recall of word forms and meanings will be tested 5 minutes after the learning session on the second day, and again one week later. After the one-week recall testing, a picture-pointing recognition task will also be completed.

In both conditions, children will initially hear the word paired with a photo (Study trial: This is a nepp. It's a nepp. A nepp likes rain.), immediately be asked to recall the word (Retrieval trial: What's this called?), and then see/hear it again (Study trial: This is a nepp. It's a nepp. A nepp likes rain.). After three other words are presented, the children will be asked to recall the original word (nepp) again (What's this called? What does it like?); this retrieval trial is followed by a study or "feedback" trial (This is a nepp. It's a nepp. A nepp likes rain.). The "3" spaced retrieval schedule will continue for the rest of the learning session. The difference between conditions is this: in the adaptive condition, if the child is unsuccessful in retrieving the word form, whether on the initial trial or on one of the "3" spaced trials, the subsequent study/feedback trial will be followed by an additional immediate retrieval trial for that word. If, on the other hand the child retrieves the word form successfully, the next retrieval - study sequence will appear after three intervening words. In the standard condition, an unsuccessful recall attempt will be followed by a study trial but there will be no additional immediate retrieval opportunity. Note that while children will also be asked to retrieve the word meaning (what it likes), unsuccessful recall of this information will not trigger an additional immediate retrieval opportunity. This is based on previous findings showing that the real difficulty for children with DLD is recalling the phonetic form of words, rather than meaning information.

The investigators predict that the strategic placement of additional immediate retrieval trials after incorrect spaced retrieval trials in the adaptive condition will increase the likelihood of the child's success on the next spaced retrieval trial. Findings show that spaced retrieval needs to be successful in order to build strength and promote long-term retention. With the boost to encoding provided by the immediate retrieval trial for words the child is having difficulty remembering, the word form may be more firmly encoded and more likely to be recalled on the spaced retrieval trials. This should lead to higher absolute levels of word learning in the adaptive condition compared to the standard condition.

ELIGIBILITY:
Inclusion Criteria:

* a significant deficit in language ability (language test score below cutoff for best sensitivity/specificity) or documented age-appropriate language ability.
* normal hearing.
* no evidence of neurological damage or disease.
* scores on tests of nonverbal intelligence above the intellectual disability range
* not within Autistic range on Autism screening test
* native English speaker (can be bilingual)

Exclusion Criteria:

* failed hearing screening
* known neurological damage or disease
* scores on tests of nonverbal intelligence below the intellectual disability range (standard score less than 75)
* autism spectrum disorder
* non-native English speaker

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Word Form Recall Accuracy (Number of Words Correctly Recalled) on Adaptive and Standard Retrieval Schedules at 5 Mins | 5 minutes after end of learning period
  5 minutes after second learning session, child is asked to recall and say the word associated with each novel referent learned under one of two conditions: one in which retrieval trials occurred on an adaptive schedule and one in which retrieval trials occurred on the standard schedule.
Word Form Recall Accuracy (Number of Words Correctly Recalled) on Adaptive and Standard Retrieval Schedules at 1 week | 1 week after end of learning period
  1 week after second learning session, child is asked to recall and say the word associated with each novel referent learned under one of two conditions: one in which retrieval trials occurred on adaptive schedule and one in which retrieval trials occurred on the standard schedule.
Word Meaning Recall Accuracy (Number of Semantic Associations Correctly Recalled) on Adaptive and Standard Retrieval Schedules at 5 Mins | 5 minutes after end of learning period
  5 minutes after second learning session, child is asked to recall and say the semantic information associated with each novel referent learned under one of two conditions: one in which retrieval trials occurred on an adaptive schedule and one in which retrieval trials occurred on the standard schedule.
Word Meaning Recall Accuracy (Number of Semantic Associations Correctly Recalled) on Adaptive and Standard Retrieval Schedules at 1 week | 1 week after end of learning period
  1 week after second learning session, child is asked to recall and say the semantic information associated with each novel referent learned under one of two conditions: one in which retrieval trials occurred on an adaptive schedule and one in which retrieval trials occurred on the standard schedule.
Word Recognition (Number of Words Accurately Identified) on on Adaptive and Standard Retrieval Schedules | 1 week after end of learning period
  Upon hearing a novel word, the child is asked to indicate (by pointing) which picture among 4 options is referred to; for words learned on the adaptive condition and for words learned on the standard condition.

SECONDARY OUTCOMES:
Standard Score on Peabody Picture Vocabulary Test, 5th Edition | at enrollment
  The Peabody Picture Vocabulary is an individually administered, norm-reference test that assesses receptive vocabulary for children and adults ages 2 years 6 months to 90 years and older. Standard scores are derived from number correct. Standard scores between 85 and 115 (1 SD above and below the mean of 100) are interpreted as reflecting receptive vocabulary levels expected for age.
Years of Maternal Education | at enrollment
  Primary care-giver provides information regarding highest academic degree attained, converted to years of education

CONTACTS AND LOCATIONS:
Overall Officials: Laurence B Leonard, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-10-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT06995014/ICF_000.pdf